CLINICAL TRIAL: NCT06135532
Title: Effect of Non-surgical Periodontal Treatment on Chemerin, Fetuin-A, IL-34 and IL-13 Levels in Type 2 Diabetic Periodontitis Patients
Brief Title: Chemerin, Fetuin-A, IL-34 and IL-13 Levels in Diabetic Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAG-A-080519-0172
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis; Diabetes Mellitus, Type 2
Keywords: periodontitis; Diabetes mellitus; periodontal therapy
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Non-Periodontitis (No Intervention): Only received instructions in proper self-performed plaque control measures, including brushing and interproximal cleaning with dental floss and interdental brushes.
- Non-Peridontitis with T2DM (No Intervention): Only received instructions in proper self-performed plaque control measures, including brushing and interproximal cleaning with dental floss and interdental brushes.
- Periodontitis (Active Comparator): The patients received instructions in proper self-performed plaque control measures, including brushing and interproximal cleaning with dental floss and interdental brushes.
  The patients underwent quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment was completed in a total of 4 sessions in four weeks.
  Interventions: Procedure: Non-Surgical Periodontal Treatment
- Periodontitis with well-controlled T2DM (Active Comparator): The patients received instructions in proper self-performed plaque control measures, including brushing and interproximal cleaning with dental floss and interdental brushes.
  The patients underwent quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment was completed in a total of 4 sessions in four weeks.
  Interventions: Procedure: Non-Surgical Periodontal Treatment
- Periodontitis with poorly-controlled T2DM (Active Comparator): The patients received instructions in proper self-performed plaque control measures, including brushing and interproximal cleaning with dental floss and interdental brushes.
  The patients underwent quadrant-wise full-mouth subgingival scaling and root planning under local anesthesia. The entire non-surgical periodontal treatment was completed in a total of 4 sessions in four weeks.
  Interventions: Procedure: Non-Surgical Periodontal Treatment

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Treatment — Nonsurgical periodontal therapy primarily aims to control microbial periodontal infection by removing bacterial biofilm, calculus, and toxins from periodontally involved root surfaces. Performing a thorough periodontal debridement under local anesthesia will stop disease progression and improve active disease's clinical signs and symptoms.
  Arms: Periodontitis; Periodontitis with poorly-controlled T2DM; Periodontitis with well-controlled T2DM

SUMMARY:
The present study aimed to assess the effect of non-surgical periodontal treatment on serum and salivary chemerin, fetuin-A, IL-34 and IL-13 levels in periodontitis with and without diabetes mellitus (DM) type 2. 22 non-periodontitis, 22 non-periodontitis with DM, 22 Stage III/IV Grade C periodontitis, 22 tage III/IV Grade C periodontitis with well-controlled DM and 22 tage III/IV Grade C periodontitis with poorly-controlled DM patients were enrolled. At baseline, serum and saliva samples were collected, and the whole mouth clinical periodontal parameters were recorded from all subjects. Periodontitis patients received non-surgical periodontal therapy. Clinical parameters were re-measured, and samples were re-collected 1 and 3 months after therapy from periodontitis patients. Serum and salivary protein levels were analyzed by ELISA. Data were analyzed using appropriate statistical tests.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) increases the risk for severe periodontal disease by three times, making it a risk factor for the progression of periodontitis. Periodontitis works as a focus of local infection and a source of low-grade chronic inflammation. Periodontal therapy primarily targets the microbial component of the disease by mechanical debridement of tooth surfaces.

Chemerin, an adipose tissue-specific adipokine, influences the glucose pathway, lipid metabolism, inflammation levels, chemotaxis of immature dendritic cells, and integration of macrophage-phagocytic activity to extracellular matrix proteins and adhesion molecules. Fetuin-A impedes insulin receptor tyrosine kinase, thus affiliated with insulin resistance, metabolic syndrome, and an increased risk for type 2 diabetes mellitus. Interleukin (IL)-34 modulates myeloid cell differentiation, proliferation, and survival. Depending on the microenvironment, IL-34 can transform circulating monocytes into specific non-resident macrophages with a "pro-inflammatory" M1 phenotype or an "anti-inflammatory" M2 phenotype. IL-13 inhibits the release of inflammatory cytokines, such as IL-1, IL-6, and TNF-α, from monocytes and macrophages.

This study is the first controlled clinical study that examines the levels of chemerin, fetuin-A, IL-34, and IL-13 in saliva and serum in periodontitis with and without T2DM (well-controlled and poorly-controlled T2DM) and evaluates the situation before and after the treatment. The first hypothesis of this study is that in periodontitis groups, chemerin and IL-34 levels will be high in saliva and serum, and IL-13 and fetuin-A levels will be low in contrast to the non-periodontitis groups. The second hypothesis of this study is that in T2DM groups, fetuin-A and chemerin levels will be high compared to participants without T2DM. The third hypothesis of this study, after periodontal treatment, chemein and IL-34 levels will decrease, and IL-13 and fetuin-A will increase in saliva and serum. Based on these hypotheses, the study aims to compare the levels of chemerin, fetuin-A, IL-34, and IL-13 in saliva and serum of nonperiodontitis controls (NP), NP with T2DM (DM.NP), periodontitis (P), P with well-controlled T2DM (WDM.P) and P with poorly-controlled T2DM (PDM.P) subjects and to evaluate the effect of periodontal treatment.

A total of 110 participants, 22 NP, 22 DM.NP, 22 P, 22 WDM.P, and 22 PDM.P were included in this study. The whole mouth clinical periodontal examination included measurement of probing depth (PPD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI), and plaque index (PI) at 6 sites per tooth, except the third molars. The presence and type of the alveolar bone loss were assessed on the digital panoramic radiograph in each participant, which was supplemented with periapical radiographs if necessary.

The periodontal status of each patient was evaluated by a single calibrated periodontist with a manual probe. The diagnosis of periodontitis or periodontally health was determined according to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions. NP individuals (healthy and gingivitis) (n=22) in the control group had no sites with PD >3 mm and CAL >2 mm and no radiographic evidence of alveolar bone loss. NP group also exhibited no history of periodontitis. The periodontitis stage III/IV patients had a minimum of three teeth apart from the first molars and incisors showing CAL ≥5 mm and PD ≥6 mm. Radiographic bone loss extending from coronal to middle third or beyond. Bone loss %/age was higher than 1.0.

The diagnosis of patients with T2DM was based on the criteria given by the World Health Organization. Both well-controlled and poorly-controlled diabetic patients, diagnosed at least one year ago as having T2DM and treated with oral anti-diabetics and/or insulin, no major diabetic complications (retinopathy, nephropathy, neuropathy), were included.

Treatment

The recruited periodontitis patients received conventional quadrant scaling and root planning (SRP) under local anesthesia in a total of 4 sessions in four weeks. SRP was performed by the same periodontist using ultrasonic inserts and manual periodontal curettes. Re-evaluations were performed at 1 and 3 months following the completion of the SRP. No periodontal intervention was carried out in the non-periodontitis controls.

Saliva and serum Sampling A total of 5 mL of unstimulated whole saliva was collected by passive drool method between 9:00 and 10:00 a.m. The participants were advised to avoid food consumption for three hours before sample collection. The participants were seated upright, and saliva was collected over 5 minutes with instructions to pool saliva in the floor of the mouth and passively drool it into a sterile glass beaker. Then, saliva samples are immediately transferred to a 2 mL polypropylene tube and stored at -80°C. A total of 10,5 mL of blood was collected from the antecubital fossa by the venepuncture method. Serum was isolated from the blood by centrifuging at 4000 rpm for 12 minutes, followed by its rapid transfer to a sterile polypropylene tube and storage at -80°C.

Biomarker Immunoassays Saliva and serum samples were thawed on ice. The saliva samples were centrifuged at 5000 rpm for 15 minutes at room temperature, and supernatants were immediately used for assays. Using commercial kits, serum and salivary samples of chemerin, fetuin-A, IL-34, and IL-13 were measured by ELISA.

Statistical Analysis Shapiro Wilk's normality test was applied to determine the clinical and biochemical data distribution. Nonparametric tests were used because the variables did not follow a normal distribution. The gender distributions among groups were analyzed using the Chi-Square test. Multiple comparisons of the clinical and biochemical parameters were analyzed using the Kruskal-Wallis; if significance occurred, the Bonferroni-adjusted Mann-Whitney U test was applied for paired comparisons. Intragroup comparisons were performed using the Wilcoxon signed-rank test. The correlations among clinical and biochemical parameters at baseline were performed using Spearman's rank correlation analysis. Multinomial logistic regression was used to determine associations between periodontitis groups and biochemical parameters. The level of significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker individuals
* having ≥20 teeth present (except third molars)
* individuals with non-periodontitis (healthy or gingivitis) and stage III grade C periodontitis diagnoses
* diagnosed at least one year ago as having T2DM and treated with oral anti-diabetics and/or insulin, no major diabetic complications (retinopathy, nephropathy, neuropathy)

Exclusion Criteria:

* having any diagnosed medical disorders other than diabetes mellitus, such as cardiovascular diseases, rheumatoid arthritis, immunological and mucocutaneous diseases
* usage of antibiotics, non-steroidal anti-inflammatory drugs, and immunosuppressive agents within the past 6 months.
* periodontal treatment within the preceding 6 months.
* pregnant/ lactating/ postmenopausal females.
* current orthodontic treatment.

Ages: 23 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
salivary chemerin level (ng/ml) | baseline to 3 months after non-surgical
  change in salivary chemerin levels
salivary fetuin-A level (ng/ml) | baseline to 3 months after non-surgical
  change in salivary fetuin-A levels
salivary IL-34 level (pg/ml) | baseline to 3 months after non-surgical
  change in salivary IL-34 levels
salivary IL-13 level (pg/ml) | baseline to 3 months after non-surgical
  change in salivary IL-13 levels

SECONDARY OUTCOMES:
serum chemerin level (ng/ml) | baseline to 3 months after non-surgical
  change in serum chemerin levels
serum fetuin-A level (ng/ml) | baseline to 3 months after non-surgical
  change in serum fetuin-A levels
serum IL-34 level (pg/ml) | baseline to 3 months after non-surgical
  change in serum IL-34 levels
serum IL-13 level (pg/ml) | baseline to 3 months after non-surgical
  change in serum IL-13 levels

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Selin Yıldırım, PhD, Principal Investigator — Department of Periodontology, Faculty of Dentistry, Marmara University, Istanbul, Turkey
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorgulu NG, Gungormek HS, Kalkan Y, Dogan B. Evaluation of chemerin, fetuin-A, interleukin-34, and interleukin-13 levels following periodontal treatment in diabetes mellitus. Clin Oral Investig. 2025 Sep 11;29(10):448. doi: 10.1007/s00784-025-06539-3. PMID 40932532